CLINICAL TRIAL: NCT04163120
Title: Effects of a Low Calorie Mediterranean Ketogenic Diet in Women With Polycystic Ovary Syndrome
Brief Title: Effects of a Ketogenic Diet on PCOS Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Palermo (Other); Universita di Verona (Other); Vita-Salute San Raffaele University (Unknown)
Responsible Party: Principal Investigator, Antonio Paoli, Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDPCOS
Record Dates: First submitted 2019-11-10; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): In this single arm study subjects follow a low calorie mediterranean ketogenci diet
  Interventions: Other: Low calorie Mediterranean ketogenic diet with phytoextracts (KEMEPHY)

INTERVENTIONS:
Other: Low calorie Mediterranean ketogenic diet with phytoextracts (KEMEPHY) — The KEMEPHY diet (24-29) is a Mediterranean low calories ketogenic protocol (about 1000/1100 Kcal/day) with the use of some phytoextracts. During this protocol subjects are allowed to eat with no limits green leafy vegetables, cruciferous, zucchini, cucumbers and eggplants. The quantity of meat, eggs and fish was limited to once a day (120g of meat or 200g of fish or 1 egg) Table 1. Moreover, subjects daily consumed four food supplements and liquid herbal extracts. Food supplements are high proteins (19g/portion) and very low carbohydrate (3.5g/portion) formulas simulating the aspect and taste of common carbohydrate rich foods added with dry phytoextracts (30). Liquid herbal extracts were used for their draining /toning activity, useful to reduce some commonly reported light side effects of ketogenic diets as constipation, headache and halitosis.

SUMMARY:
The aim of the study is to investigate the effects of a low calorie Mediterranean ketogenic diet on Polycystic Ovary Syndrome (PCOS) related outcomes.

DETAILED DESCRIPTION:
Fourteen overweight women with diagnosis of Polycystic Ovary Syndrome (PCOS) will undergo to a low calorie ketogenic Mediterranean diet with phyoextracts (KEMEPHY) for 12 week. Changes in body weight, body mass index (BMI), fat body mass (FBM), lean body mass (LBM), visceral adipose tissue (VAT), insulin, glucose, HOMA-IR, total cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL(, triglycerides (TGs), total and free testosterone, luteinizing hormone (LH), follicle stimulating hormone (FSH); dehydroepiandrosterone sulfate (DHEAs), estradiol, progesterone, sex hormone binding globulin (SHBG) and Ferriman Gallwey score will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of PCOS according Rotterdam Criteria (at least 2 of 3 between

* oligo/anovulation
* hyperandrogenism
* clinical (hirsutism or less commonly male pattern alopecia) or biochemical (raised FAI or free testosterone) polycystic ovaries on ultrasound Other inclusion criteria
* fertile age (18-45 years);
* BMI> 25 kg/m2,
* desire to lose weight;
* acceptance not to use contraceptives during the experimental period

Exclusion Criteria:

* pregnancy and lactation,
* hormonal therapy and/or insulin-sensitizers in the last 2 months,
* hepatic, renal and heart diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks
  Body weight will be measured by an electronic scale
Fat body mass | 12 weeks
  will be analysed by Dual X Ray Absorptiometry (DEXA) Hologic HorizonTM QDR RSeries Bedford, Massachusetts, USA
LH | after 12 weeks
  LH will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
FSH | 12 weeks
  FSH will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
Total testosterone | 12 weeks
  Total testosterone will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
Insulin | 12 weeks
  Insulin will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
DHEAS | 12 weeks
  DHEAS will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
progesterone | 12 weeks
  progesterone will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
estradiol | 12 weeks
  estradiol will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
SHBG | 12 weeks
  SHBG will be measured by immunochemiluminescent method (Roche Cobas e601, Roche Diagnostics, Mannheim, Germany)
HOMA | 12 weeks
  HOMA-IR will be calculated according to the formula "insulinemia (μU/mL) x glycemia (mmol/L)/22.5
blood glucose | 12 weeks
  blood glucose will be measured by enzymatic method with esokinase (Roche Cobas e702, Roche Diagnostics, Mannheim, Germany)
Hirsutism . | 12 weeks
  we will use Ferriman Gallwey Score. A score of 1 to 4 is given for nine areas of the body. A total score less than 8 is considered normal, a score of 8 to 15 indicates mild hirsutism, and a score greater than 15 indicates moderate or severe hirsutism. A score of 0 indicates absence of terminal hair.

SECONDARY OUTCOMES:
Ketone bodies | 12 weeks
  Ketone bodies will be measured by Precision Xtra® Blood β-Ketone Test Strips and Precision Xtra® (28) (Abbott Laboratories, Illinois 60064-3500, USA)
total cholesterol | 12 weeks
  total cholesterol will be measured by enzymatic colorimetric in homogenous phase (Roche Cobas e702, Roche Diagnostics, Mannheim, Germany)
HDL cholesterol | 12 weeks
  HDL cholesterol will be measured by enzymatic colorimetric in homogenous phase (Roche Cobas e702, Roche Diagnostics, Mannheim, Germany)
LDL cholesterol | 12 weeks
  LDL cholesterol will be measured by enzymatic colorimetric in homogenous phase (Roche Cobas e702, Roche Diagnostics, Mannheim, Germany)
Triglycerides | 12 weeks
  TGs by an enzymatic colorimetric method (Roche Cobas e702, Roche Diagnostics, Mannheim, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paoli A, Grimaldi K, Toniolo L, Canato M, Bianco A, Fratter A. Nutrition and acne: therapeutic potential of ketogenic diets. Skin Pharmacol Physiol. 2012;25(3):111-7. doi: 10.1159/000336404. Epub 2012 Feb 11. PMID 22327146
- [Background] Paoli A, Rubini A, Volek JS, Grimaldi KA. Beyond weight loss: a review of the therapeutic uses of very-low-carbohydrate (ketogenic) diets. Eur J Clin Nutr. 2013 Aug;67(8):789-96. doi: 10.1038/ejcn.2013.116. Epub 2013 Jun 26. PMID 23801097
- [Background] Paoli A, Mancin L, Bianco A, Thomas E, Mota JF, Piccini F. Ketogenic Diet and Microbiota: Friends or Enemies? Genes (Basel). 2019 Jul 15;10(7):534. doi: 10.3390/genes10070534. PMID 31311141
- [Background] Mavropoulos JC, Yancy WS, Hepburn J, Westman EC. The effects of a low-carbohydrate, ketogenic diet on the polycystic ovary syndrome: a pilot study. Nutr Metab (Lond). 2005 Dec 16;2:35. doi: 10.1186/1743-7075-2-35. PMID 16359551
- [Background] Galletly C, Moran L, Noakes M, Clifton P, Tomlinson L, Norman R. Psychological benefits of a high-protein, low-carbohydrate diet in obese women with polycystic ovary syndrome--a pilot study. Appetite. 2007 Nov;49(3):590-3. doi: 10.1016/j.appet.2007.03.222. Epub 2007 Apr 4. PMID 17509728
- [Derived] Moro T, Monaco L, Naro F, Reggiani C, Paoli A. Exercise Intensity and Rest Intervals Effects on Intracellular Signals and Anabolic Response of Skeletal Muscle to Resistance Training. J Strength Cond Res. 2024 Oct 1;38(10):1695-1703. doi: 10.1519/JSC.0000000000004209. Epub 2022 Jan 5. PMID 40168063
- [Derived] Paoli A, Mancin L, Giacona MC, Bianco A, Caprio M. Effects of a ketogenic diet in overweight women with polycystic ovary syndrome. J Transl Med. 2020 Feb 27;18(1):104. doi: 10.1186/s12967-020-02277-0. PMID 32103756